CLINICAL TRIAL: NCT05209555
Title: Observational Study on the Predictive Value of the BAMCOG and Cortisol Levels for the Incidence of Postoperative Delirium/Postoperative Acute Encephalopathy Measured by the MoCA and the DeltaScan in Patients Who Undergo Aortic Valve Replacement Surgery
Brief Title: Preoperative BAMCOG and Cortisol and Postoperative DeltaScan in AVR Patients (Aortic Valve Replacement)
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Mariska te Pas, Principal Investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: CZE-2021.57
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Delirium; Cognitive Impairment; Cognitive Dysfunction; Cognitive Dysfunction, Postoperative; Delirium in Old Age; Postoperative Delirium
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MoCA — MoCA test to identify Mild Cognitive Impairment
Device: BAMCOG — Three games, compared to the MoCA to identify Mild Cognitive Impairment
Diagnostic Test: DeltaScan — EEG to detect acute encephalopathy
Diagnostic Test: Salivette — To collect saliva for cortisol analysis
Diagnostic Test: Pilocarpine iontophoresis — To collect sweat for cortisol analysis

SUMMARY:
There is lack of attention to preoperative cognitive function and delirium in elderly who underwent surgery. The investigators are investigating different tools that can help to screen for cognitive dysfunction and delirium in the future.

DETAILED DESCRIPTION:
Background of the study:

The mean age of surgical patients is rising worldwide and this is associated with more multi-morbidity. Especially geriatric patients who undergo surgery have a higher risk to develop Postoperative Cognitive Dysfunction or a Postoperative Delirium, which leads to higher morbidity and mortality after surgery and this leads to higher healthcare costs.

A delirium is an acutely disturbed state of mind characterized by restlessness, illusions, and incoherence, occurring in intoxication, fever, and other disorders and can fluctuate over time. The hypoactive delirium, the most common type of delirium, is hard to recognize compared to the active delirium that is expressed by restlessness and agitation.

Postoperative cognitive dysfunction is defined as a new cognitive impairment arising after a surgical procedure. Its diagnosis requires both pre- and postoperative psychometric testing. Its manifestations are subtle and manifold, depending on the particular cognitive domains that are affected, and therefore hard to recognize too.

To assess preoperative cognitive function in large groups of patients, it's needed to have a simple and quick tool to screen. In this study, the investigators use the BAMCOG, which is a tool with 3 short games played on a tablet that can provide information about cognitive functioning. When writing this new study protocol, a validation study in which the BAMCOG is validated against the MoCA is running.

Beside the BAMCOG, another instrument will be investigated. The DeltaScan is an EEG delta waves measurement to identify patients with a (hypoactive) delirium. Delta waves are slow brainwaves that have been seen in sedated patients and even inpatients with an active or hypoactive delirium. A study of Kimchi et al. studied whether routine clinical EEG findings, including slowing, are correlated with delirium severity in a heterogeneous population with various causes of altered mental status and found that generalized slowing on routine clinical EEG strongly correlates with delirium and may be a valuable biomarker for delirium severity (OR 7.4, 95% CI 3.8-14.4).

A lot remains unclear about the biological mechanisms in the development of a delirium after surgery, although in literature are directions that inflammatory reactions and the neuro-endocrine system play an important role. That is the reason for investigating the relation between cortisol levels in blood, saliva and sweat and the development of postoperative acute encephalopathy.

Objective of the study:

1. The predictive value of the BAMCOG for developing postoperative delirium/postoperative acute encephalopathy in patients who underwent AVR surgery
2. Concurrent validation of the BAMCOG with the MoCA
3. The relation between cortisol levels in blood, saliva and sweat and the development of postoperative delirium/postoperative acute encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* age >65 year
* scheduled for AVR surgery
* Able to play the BAMCOG games after instruction
* (Near) native (dutch)

Exclusion Criteria:

* mental disorder
* learning disorder
* diagnosed dementia at start of study
* alcohol abuses
* lithium/clozapine use because of DeltaScan
* sedation/RASS -4/-5 because of DeltaScan
* not able to sign informed consent
* implanted pacemaker, defibrillator or neurostimulator because of pilocarpine iontophoresis
* history of insults
* pregnant women
* allergy to pilocarpine
* damaged skin (forearm)

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 50 patients 65 years or older who will undergo AVR-bio surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Prognostic value of the preoperative BAMCOG to predict postoperative delirium | BAMCOG and DeltaScan - preoperative 1 day, postoperative day 1, 3, 7.

SECONDARY OUTCOMES:
Correlation BAMCOG scores and MoCA scores | MoCA - preoperative 1 day, postoperative day 1, 3, 7
Prognostic value of cortisol measures (Sweat, Saliva, Serum) to predict postoperative delirium | Preoperative at home and postoperative day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No